CLINICAL TRIAL: NCT02736604
Title: Evaluation of Impact of Nitrous Oxide on PONV in Breast Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Vijaya P Patil, professor and Anaesthetist, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: project number 1650
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Laryngeal Masks; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air anesthesia (Experimental): air will be used as carrier agent for maintenance of anesthesia
  Interventions: Drug: air anesthesia; Device: laryngeal mask airway (LMA Supreme Size 3/4; Drug: sevoflurane
- Nitrous Oxide anesthesia (Active Comparator): nitrous oxide will be used as carrier agent for maintenance of anesthesia
  Interventions: Drug: nitrous oxide anesthesia; Device: laryngeal mask airway (LMA Supreme Size 3/4; Drug: sevoflurane

INTERVENTIONS:
Drug: nitrous oxide anesthesia — General anesthesia will be maintained by 40% oxygen (FiO2 0.4) with Nitrous Oxide and volatile anesthetic sevoflurane through laryngeal mask airway (LMA Supreme Size 3/4) or endotracheal tube (Size 7.0-7.5). All patients will receive standard anesthetic care and monitoring
  Arms: Nitrous Oxide anesthesia
Drug: air anesthesia — General anesthesia will be maintained by 40% oxygen (FiO2 0.4) with air and volatile anesthetic sevoflurane through laryngeal mask airway (LMA Supreme Size 3/4) or endotracheal tube (Size 7.0-7.5). All patients will receive standard anesthetic care and monitoring
  Arms: Air anesthesia
Device: laryngeal mask airway (LMA Supreme Size 3/4
Drug: sevoflurane

SUMMARY:
Postoperative nausea and vomiting (PONV) is considered one of the most unpleasant postoperative discomforts and lead to serious complications of aspiration of gastric contents, suture dehiscence, esophageal rupture, subcutaneous emphysema, or pneumothorax. The incidence of PONV is 30-40% in normal population and touches a peak of 75-80% in certain high-risk groups. PONV is associated with delayed recovery and prolonged hospital stay and is associated with significant morbidity. It may also result in delayed discharge, which is particularly significant after potentially ambulatory surgery. Women are 2 to 3 times more susceptible to PONV than men and breast surgery, which is primarily done in an outpatient setting, is associated with high incidence of PONV, ranging between 15% and 84% in the absence of prophylactic treatment.

Nitrous oxide (N2O) has analgesic and sedative properties but may potentially increase the incidence of PONV. N2O might increase the incidence of PONV by several potential mechanisms: (1) increase in middle ear pressure (2) bowel distension, (3) activation of the dopaminergic system in the chemoreceptor trigger zone and (4) interaction with opioid receptors. N2O has been demonstrated to increase the incidence of PONV in some studies but not in others. The present study is undertaken to evaluate the effect of nitrous oxide- free general anesthesia on the undesirable clinical outcome of PONV.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I and II female patients aged 18 years or over posted for Breast Surgeries under General Anesthesia in the main operating rooms

Exclusion Criteria:

1. ASA III, IV, V female patients
2. Age less than 18 years
3. Patients undergoing Breast Reconstructive Surgery
4. Patients with contraindications to Fentanyl, Diclofenac, Paracetamol, Atracurium
5. Chronic pain patients on long-term opioid medication
6. Use of regional anesthetic technique (e.g. Paravertebral Block)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
incidence and severity of post operative nausea and vomiting | up to 24 hours after surgery
  Patients will be followed for 24 hours post-surgery or discharge from hospital whichever is earlier. postoperative nausea and vomiting intensity scale will be used to assess incidence and severity of nausea and vomiting.

SECONDARY OUTCOMES:
measurement of pain score and analgesic requirements | up to 24 hours after surgery
  Patients will be followed for 24 hours post-surgery or discharge from hospital whichever is earlier. Pain score will be measured by Visual Analogue Scale from 0-10.
Airway device cuff pressures | During the surgery
  airway device cuff pressure will be measured during the surgery either endotracheal tube or laryngeal mask airway which ever is applicable

CONTACTS AND LOCATIONS:
Overall Officials: vijaya p patil, MD, Principal Investigator — Department of Anaesthesia, Critical Care and Pain, Tata Memorial Hospital, parel, mumbai, India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes